CLINICAL TRIAL: NCT01887054
Title: Effect of Visuospatial Training Tasks on Freezing of Gait in Parkinson's Disease
Brief Title: Freezing of Gait in Parkinson's Disease
Acronym: FOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00045495
Record Dates: First submitted 2013-06-19; First posted 2013-06-26 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Training Group (Active Comparator): There are 2 study visits. Subjects in this group will complete the following:
  Visit 1
  * Gait evaluation
  * Neuropsychological testing
  * Questionnaires and assessments
  * Taught how to complete a visual problem-solving task (Tower of Hanoi)
  * Given a diary to record training at home.
  In-home
  •For 6 weeks at home, complete the in-home visual problem-solving tasks as instructed at Visit 1
  Visit 2
  * Gait evaluation
  * Neuropsychological testing
  * Questionnaires and assessments
  Interventions: Device: Tower of Hanoi
- Non Training Group (Placebo Comparator): There are 2 study visits. Subjects in this group will complete the following:
  Visit 1
  * Gait evaluation
  * Neuropsychological testing
  * Questionnaires and assessments
  Visit 2
  * Gait evaluation
  * Neuropsychological testing
  * Questionnaires and assessments
  Interventions: Other: Placebo group - non use of Tower of Hanoi

INTERVENTIONS:
Device: Tower of Hanoi
  Arms: Training Group
Other: Placebo group - non use of Tower of Hanoi
  Arms: Non Training Group

SUMMARY:
This study is designed to evaluate whether a specific visuospatial training task will change gait performance of Parkinson's disease (PD) patients in doorways, specifically freezing of gait.

DETAILED DESCRIPTION:
This study is a randomized, prospective, single-blinded six-week study in PD patients with freezing of gait (FOG).

This study will involve 2 study groups:

Group A - training group; Group B - no training group/controls.

Both groups will complete a gait evaluation and neuropsychological testing. Group A will also practice an in-home visuospatial task for 30 minutes, 4-6 days per week for six weeks. Group B will not complete the in-home tasks.

Participation in this study is expected to last 6-8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: greater than 18 years old and without an upper age limit
* diagnosis of idiopathic PD exhibiting at least 2 or 3 cardinal signs (bradykinesia, rigidity, and resting tremor)
* Ambulate independently without an assistive device for at least 60 meters
* Freezing of gait episodes confirmed through the FOG-Q and evaluation by a fellowship trained Movement Disorder neurologist
* Willingness and ability to participate in training and complete training diary
* Documented FOG-Q and Unified Parkinson's Disease Rating Scale (UPDRS) II
* Ability to sign informed consent
* Pregnant females will be included in the study and there are no known risks to the pregnant female or fetus

Exclusion Criteria:

* Inability to complete questionnaires
* Unwillingness to participate in training, complete all questionnaires and training diary
* Subjects with secondary causes of parkinsonism
* Significant dementia (MOCA <20)
* Prior deep brain stimulation (DBS) surgery or pallidotomy
* Subjects cannot participate in any form of Physical Therapy, Occupational Therapy or Speech Therapy during the study period
* Subjects cannot start any new medications during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Double Limb Support (DLS) | 6 weeks
  Primary outcome will be the percent of the gait cycle spent in DLS. This will be evaluated using a GaitRite via a continuous walk, with subjects walking an 18-20 meter oval loop three times continuously.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stacy, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States